CLINICAL TRIAL: NCT01098279
Title: Multidisciplinary Approach to the Study of Chronic Pelvic Pain: Trans-MAPP Epidemiology and Phenotyping (EP) Study
Brief Title: Chronic Pelvic Pain Study of Individuals With Diagnoses or Symptoms of Interstitial Cystitis and/ or Chronic Prostatitis
Acronym: MAPP-EP
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 810643; U01DK082316 (NIH)
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Interstitial Cystitis; Chronic Prostatitis
Keywords: Interstitial Cystitis; Chronic Prostatitis; Urological Chronic Pelvic Pain; Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA Blood Urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Multidisciplinary Approach to the Study of Chronic Pelvic Pain (MAPP) Research Network has been established to focus on a broader approach to the study of Interstitial Cystitis (IC)/Painful Bladder Syndrome (PBS) in men and women, and Chronic Prostatitis (CP)/Chronic Pelvic Pain Syndrome (CPPS) in men, than previously undertaken. Participants with some form or symptoms of IC or CP are being asked to join the Trans-MAPP Epidemiology and Phenotyping (EP) Study.

As with many chronic pain disorders, IC and CP are poorly understood, and treatment is often not helpful. The goal of this study is to better understand how pain is felt in people with IC or CP. The MAPP EP Study is an observational study that will enroll approximately 360 participants from 6 Discovery Sites and 3 Satellite Sites across the U.S. We will ask questions and gather information about the health and life of the participants for research purposes. No study treatment or interventions will be given to participants in MAPP. We hope that this study will lead to improvement in the treatment of IC and CP.

DETAILED DESCRIPTION:
Potentially eligible participants will be scheduled for an eligibility screening session, followed by an extensive baseline phenotyping session, which together are expected to take approximately 2.5 hours to complete. Participants will be provided with breaks as needed during the clinic visit. The eligibility screening session is intended to collect the minimally sufficient data to confirm eligibility, so that the extensive baseline phenotyping session is initiated only for participants highly likely to be confirmed after the 48 hour urine culture results are known.

Participants who enroll in the study and complete a baseline clinic visit will be followed up with bi-weekly and bi-monthly internet-based questionnaires, as well as in-clinic visits at 6 and 12 months.

Participants will provide self-reported symptom data using web based internet tools on a bi-weekly basis. These questions are expected to be completed within 5-7 minutes.

A more extensive set of questionnaires will be administered to each participant every two months during the 12-month study period. The bi-monthly assessment will also be administered via the internet, and the questions are expected to be completed within 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible for the Trans-MAPP EP if they meet the following:

1. Participant has signed and dated the appropriate Informed Consent document.
2. Agreed to participate in Trans-MAPP EP Study procedures.
3. Participant reports a response of at least 1 on the pain, pressure or discomfort scale.

For males or females (IC/PBS criteria)

1. Participant reports an unpleasant sensation of pain, pressure or discomfort, perceived to be related to the bladder and/or pelvic region, associated with lower urinary tract symptoms for the majority of the time during any 3 months in the previous 6 months or for the majority of the time during the most recent 3 months.

For males only (CP/CPPS criteria)

1. Male participant reports pain or discomfort in any of the 8 domains of the Male Genitourinary Pain Index for the majority of the time during any 3 months in the previous 6 months

Exclusion Criteria:

Individuals will not be eligible for enrollment in the Trans-MAPP EP Study if they meet any of the criteria listed below. Participants who develop any of these exclusion criteria during the follow-up phase of the study will continue to be followed, and included in the cohort study.

1. Participant has an on-going symptomatic urethral stricture.
2. Participant has an on-going neurological disease or disorder affecting the bladder or bowel fistula.
3. Participant has a history of cystitis caused by tuberculosis, radiation therapy or Cytoxan/cyclophosphamide therapy.
4. Participant has augmentation cystoplasty or cystectomy.
5. Participant has a systemic autoimmune disorder (such as Crohn's Disease or Ulcerative Colitis, Lupus, Rheumatoid Arthritis, or Multiple Sclerosis).
6. Participant has a history of cancer (with the exception of skin cancer).
7. Participant has current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, etc).
8. Participant has severe cardiac, pulmonary, renal, or hepatic disease that in the judgment of the study physician would preclude participation in this study.

Exclusion Criteria for Males Only

1. Male Participant diagnosed with unilateral orchalgia, without pelvic symptoms.
2. Male Participant has a history of transurethral microwave thermotherapy (TUMT), transurethral needle ablation (TUNA), balloon dilation, prostate cryo-surgery, or laser procedure.

Exclusion Criteria for Females Only

1. Female Participant has a history of High-Grade Squamous Intraepithelial Lesion (HGSIL) / high-grade cervical dysplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Trans-MAPP EP Study population will include adult participants, at least 18 years of age, with urological chronic pelvic pain syndromes. Approximately half of the participants will be male, and half will have recent onset (within two years) of pelvic pain symptoms and/or limited treatment as determined by self-report.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Longitudinal outcomes for MAPP Participants | Baseline/6 month/12 month/ bi-weekly/bi-monthly
  Extensive data on risk factors and outcomes measures will be collected for the Trans-MAPP EP Study. These measures can be classified into a number of primary domains as described below.
  1. Single point in time: this includes measures that do not change over time, such as demographic information, "trait measures" (e.g., personality), and early life history measures. In general, these measures are collected at the initial in-person clinic visit, although some are collected in the second (6-month) in-person visit to reduce participant burden at baseline;
  2. Baseline, 6-month and 12-month phenotyping in-clinic visits;
  3. Bi-monthly personal internet-based assessment;
  4. Bi-weekly personal internet-based assessment.

CONTACTS AND LOCATIONS:
Overall Officials: J. Quentin Clemens, MD, Study Chair — University of Michigan; Christopher Mullins, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Harte SE, Schrepf A, Gallop R, Kruger GH, Lai HHH, Sutcliffe S, Halvorson M, Ichesco E, Naliboff BD, Afari N, Harris RE, Farrar JT, Tu F, Landis JR, Clauw DJ; MAPP Research Network. Quantitative assessment of nonpelvic pressure pain sensitivity in urologic chronic pelvic pain syndrome: a MAPP Research Network study. Pain. 2019 Jun;160(6):1270-1280. doi: 10.1097/j.pain.0000000000001505. PMID 31050659
- [Derived] Rodriguez LV, Stephens AJ, Clemens JQ, Buchwald D, Yang C, Lai HH, Krieger JN, Newcomb C, Bradley CS, Naliboff B; MAPP Research Network. Symptom Duration in Patients With Urologic Chronic Pelvic Pain Syndrome is not Associated With Pain Severity, Nonurologic Syndromes and Mental Health Symptoms: A Multidisciplinary Approach to the Study of Chronic Pelvic Pain Network Study. Urology. 2019 Feb;124:14-22. doi: 10.1016/j.urology.2018.11.015. Epub 2018 Nov 16. PMID 30452963
- [Derived] Schrepf A, Naliboff B, Williams DA, Stephens-Shields AJ, Landis JR, Gupta A, Mayer E, Rodriguez LV, Lai H, Luo Y, Bradley C, Kreder K, Lutgendorf SK; MAPP Research Network. Adverse Childhood Experiences and Symptoms of Urologic Chronic Pelvic Pain Syndrome: A Multidisciplinary Approach to the Study of Chronic Pelvic Pain Research Network Study. Ann Behav Med. 2018 Sep 13;52(10):865-877. doi: 10.1093/abm/kax060. PMID 30212850
- [Derived] Landis JR, Williams DA, Lucia MS, Clauw DJ, Naliboff BD, Robinson NA, van Bokhoven A, Sutcliffe S, Schaeffer AJ, Rodriguez LV, Mayer EA, Lai HH, Krieger JN, Kreder KJ, Afari N, Andriole GL, Bradley CS, Griffith JW, Klumpp DJ, Hong BA, Lutgendorf SK, Buchwald D, Yang CC, Mackey S, Pontari MA, Hanno P, Kusek JW, Mullins C, Clemens JQ; MAPP Research Network Study Group. The MAPP research network: design, patient characterization and operations. BMC Urol. 2014 Aug 1;14:58. doi: 10.1186/1471-2490-14-58. PMID 25085119
- [Derived] Clemens JQ, Mullins C, Kusek JW, Kirkali Z, Mayer EA, Rodriguez LV, Klumpp DJ, Schaeffer AJ, Kreder KJ, Buchwald D, Andriole GL, Lucia MS, Landis JR, Clauw DJ; MAPP Research Network Study Group. The MAPP research network: a novel study of urologic chronic pelvic pain syndromes. BMC Urol. 2014 Aug 1;14:57. doi: 10.1186/1471-2490-14-57. PMID 25085007
- See also: MAPP Research Network Website — http://mappnetwork.org